CLINICAL TRIAL: NCT06831994
Title: Digital Implementation of the German S3 Clinical Practice Guideline for Primary Care of Older Patients With Multimorbidity - a Cluster-randomised Clinical Evaluation Study (Gp-multitool.de)
Brief Title: Digital Implementation of the German S3 Clinical Practice Guideline for Multimorbidity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01GY2109
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Asthma Bronchiale; Breast Neoplasms; Coronary Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Pulmonary Disease, Chronic Obstructive; Obesity; Heart Failure; Chronic Low-back Pain; Depression; Osteoporosis; Rheumatoid Arthritis; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Breast Neoplasms; Coronary Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Pulmonary Disease, Chronic Obstructive; Obesity; Heart Failure; Depression; Osteoporosis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The project staff conducting patient interviews will be blinded regarding allocation of the patient's practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Care as usual
- Intervention group (Experimental): GPs in the intervention arm have to use the web application gp-multitool.de. For every participating patient they have to use at least four specific questionnaires in the first six intervention months, i.e. 1a is required, and either 2a or 2b, and either 3a or 3b, and either 4a or 4b or 4c. In the following six intervention months, GPs in the intervention arm also have to use at least four specific questionnaires, i.e., 1a is required again, and either 2a or 2b, and either 3a or 3b, and either 4a or 4b or 4c. Results from the questionnaires need to be discussed between GPs and patients. Additionally, at least one medication review during the first six intervention months is obligatory.
  Interventions: Other: gp-multitool.de

INTERVENTIONS:
Other: gp-multitool.de — The intervention is based on the digital tool gp-multitool.de. The GPs can send questionnaires by email to patients and patients can fill out questionnaires at their home or in the waiting room of the practice using any digital device with browser and access to the internet. The digital tool also includes instructions for conducting a medication review. Results will be available from the computers of attending GPs. Decisions from talks between GPs and patients can be documented in the tool. The tool includes ten questionnaires:
  1. patient preferences (including a. treatment goals, and b. involvement of other persons in decision making);
  2. social life (including a. activities and participation, and b. social support);
  3. treatment situation (including a. problems with medication, and b. treatment burden);
  4. health complaints (including a. pain, b. psychiatric disorders, and c. other complaints).
  5. resilience and protective behavior against heat.
  Arms: Intervention group

SUMMARY:
The web application gp-multitool.de is a digital tool for implementing the German S3 clinical practice guideline for multimorbidity of the German Society of General Practitioners and Family Physicians in primary care. The tool enhances evidence-based and patient-centered care by assessing and providing information relevant for the primary care of this patient group. This cluster-randomised clinical evaluation study examines the effectiveness of an intervention based on gp-multitool.de in general practitioner (GP) practices in Germany.

DETAILED DESCRIPTION:
The web application gp-multitool.de study is a digital tool for implementing the German S3 clinical practice guideline for multimorbidity of the German Society of General Practitioners and Family Physicians in primary care. The tool enhances evidence-based and patient-centered care for patients with multimorbidity by assessing and providing information relevant for the primary care of this patient group. The study intervention is based on this digital tool and aims to reduce the probability of hospital admissions (primary outcome) and their outpatient health care use, and to improve process quality of care, patients' health-related quality of life, and patient satisfaction (secondary outcomes).

This cluster-randomized clinical evaluation study examines the effectiveness of the gp-multitool.de intervention in GP practices. GPs in the intervention group implement the intervention in consultations with participating patients for 12 months. Intervention GPs gain access to the digital tool, and get a brief introduction to its functionalities, a video tutorial, a written manual, and contact data of telephone support, which can be called in case of any technical or organizational problems in relation to the digital tool. In addition, they receive a short training in the intervention and a checklist of requirements defined in the study protocol. Moreover, each intervention practice will be provided with a mobile device, facilitating inclusion of patients without access to the internet. GPs in the control group receive no intervention and provide care as usual.

Patients will be recruited from GP practices in urban and rural administrative districts in Germany. The evaluation study is based on telephone interviews of patients and their GPs. Practices will be randomized after the baseline assessment by an independent statistician who does not have access to the assessed patient and practice data. The primary outcome will be analyzed using a multilevel mixed-effects logistic regression model, and secondary outcomes will be analyzed by multilevel mixed-effects linear and negative-binomial regression models. The project staff conducting patient interviews will be blinded regarding allocation of the patient's practices.

ELIGIBILITY:
Inclusion Criteria:

* participation in a disease management program (DMP); in Germany, DMPs have been implemented in outpatient care for asthma, breast neoplasms, coronary heart disease, diabetes mellitus type 1, diabetes mellitus type 2, chronic obstructive pulmonary disease, obesity, heart failure, chronic low back pain, depression, osteoporosis, rheumatoid arthritis
* at least two of the following coexisting conditions: Hypertension, Lipid metabolism disorders, Chronic low back pain, Severe vision reduction, Joint arthrosis, Diabetes mellitus, Chronic ischemic heart disease, Thyroid dysfunction, Cardiac arrhythmias, Obesity, Hyperuricemia/Gout, Prostatic hyperplasia, Lower limb varicosis, Liver diseases, Depression, Asthma/Chronic obstructive pulmonary disease, Gynaecological problems, Atherosclerosis/Peripheral arterial occlusive disease, Osteoporosis, Renal insufficiency, Cerebral ischemia/Chronic stroke, Cardiac insufficiency, Severe hearing loss, Chronic cholecystitis/Gallstones, Somatoform disorders, Hemorrhoids, Intestinal diverticulosis, Rheumatoid arthritis/Chronic polyarthritis, Cardiac valve disorders, Neuropathies, Dizziness, Dementias, Urinary incontinence, Urinary tract calculi, Anemias, Anxiety, Psoriasis, Migraine/chronic headache, Parkinson's disease, Cancers, Allergies, Chronic gastritis/Gastroesophageal reflux disease, Sexual dysfunction, Insomnia, Tobacco abuse, Hypotension

Exclusion Criteria:

* no capacity to consent
* functional limitations precluding participation in the intervention (eg, loss of vision)
* functional limitations precluding participation in telephone interviews (eg, loss of hearing)
* limited German language skills precluding participation in telephone interviews
* participation in other trials during the observation time of the evaluation study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Whether patients have stayed at least once for at least one night in hospital during the preceding twelve months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by a standardised questionnaire. The patients will be asked how often they had been in hospital during the preceding twelve months and how long these stays had lasted. Before analysis, the outcome will be dichotomised.

SECONDARY OUTCOMES:
The number of contacts with the GP during the preceding twelve months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had visited their GP during the preceding twelve months.
The number of contacts with outpatient specialists during the preceding twelve months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had visited outpatient specialists during the preceding twelve months.
Quality of care as assessed by the summary score of the "GP-reported core set of quality indicators for older adults with multimorbidity in primary care" during the preceding twelve months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "GP-reported core set of quality indicators for older adults with multimorbidity in primary care" (Schäfer I et al. 2023, digital object identifier (DOI): https://doi.org/10.1186/s12916-023-02856-0), which has a possible range between 0 and 12 points. Higher scores indicate a better quality of primary care.
Quality of care as assessed by the summary score of the "patient-reported core set of quality indicators for older adults with multimorbidity in primary care" during the preceding twelve months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "Patient-reported core set of quality indicators for older adults with multimorbidity in primary care" (Schäfer I et al. 2023, DOI: https://doi.org/10.1186/s12916-023-02856-0), which has a possible range between 0 and 7 points. Higher scores indicate a better quality of primary care.
Self-rated health as assessed by the EuroQoL visual analogue scale | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the EuroQoL visual analogue scale (Herdman M et al. 2011, DOI: 10.1007/s11136-011-9903-x), which has a possible range between 0 and 100 points. Higher scores indicate a better self-rated health.
Health-related quality of life as assessed by the "Short-Form-Health Survey (SF-12)" questionnaire | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "Short-Form-Health Survey (SF-12)" questionnaire (Wirtz M.A. et al. 2018, DOI: 10.1026/0012-1924/a000205), which has a possible range between 0 and 100 points. Higher scores indicate a better health-related quality of life.
Patient satisfaction with chronic illness care assessed by the "Patient Assessment of Chronic Illness Care (PACIC 5A)" questionnaire | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "PACIC 5A" questionnaire (Rosemann T et al. 2007, DOI: 10.1111/j.1365-2753.2007.00786.x), which has a possible range between 1 and 5 points. Higher scores indicate a higher patient satisfaction with chronic illness care from patient's perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Schäfer, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be included in the publication as supplementary file.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available at the time of publication. No time limit is planned.
Access Criteria: No restrictions.

REFERENCES:
- [Derived] Schafer I, Menzel A, Lezius S, Krause L, Zapf A, Luhmann D, Scherer M, Paucke V, Nothacker J. Effects of a digital tool implementing the German S3 clinical practice guideline for multimorbidity in primary care (gp-multitool.de): study protocol for a cluster-randomised controlled trial. BMJ Open. 2025 Aug 3;15(8):e102086. doi: 10.1136/bmjopen-2025-102086. PMID 40754332